CLINICAL TRIAL: NCT02669329
Title: CoolSculpting the Upper Arm Using a Vacuum Applicator
Brief Title: CoolSculpting the Upper Arm Study
Acronym: ARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA15-005
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-08

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Upper arm treatment with vacuum applicator (Experimental): Subjects with clearly visible fat sufficient for treatment received bilateral CoolSculpting treatments, 1 treatment on each arm.
  Interventions: Device: CoolSculpting device with vacuum applicator.

INTERVENTIONS:
Device: CoolSculpting device with vacuum applicator. — The CoolSculpting device with a vacuum applicator will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of the ZELTIQ CoolSculpting System using a specialized surface applicator for non-invasive subcutaneous fat reduction in the upper arm.

DETAILED DESCRIPTION:
This multi-center trial will evaluate the Zeltiq CoolSculpting treatment to perform treatments in the upper arm for the reduction subcutaneous fat reduction.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat sufficient for treatment on the upper arm, which in the investigator's opinion, may benefit from the treatment.
* No weight change exceeding 5% in the preceding month.
* Subject agrees to maintain his/her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.), or implants in or adjacent to the area of intended treatment.
* History of prior surgery in the arms.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* History of carpal tunnel syndrome, compartment syndrome or deep vein thrombosis in the upper extremities.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars, infection, in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 5 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of any other unapproved investigational drug or device. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dr. Jean Carruthers Cosmetic Surgery Inc., Vancouver, British Columbia
  - Pacific Dermaesthetics, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carruthers JD, Humphrey S, Rivers JK. Cryolipolysis for Reduction of Arm Fat: Safety and Efficacy of a Prototype CoolCup Applicator With Flat Contour. Dermatol Surg. 2017 Jul;43(7):940-949. doi: 10.1097/DSS.0000000000001134. PMID 28595246

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: arms
Groups:
- Upper Arm Treatment Group: Each subject in the arm received bilateral treatment with the CoolSculpting device. Each arm was treated once.
Period: Overall Study
Arm/Group | Upper Arm Treatment Group
Started | 30; 60 arms
Completed | 30; 60 arms
Not Completed | 0; 0 arms

BASELINE CHARACTERISTICS:
Groups:
- Upper Arm Treatment With Vacuum Applicator: The CoolSculpting device with vacuum applicator will be used to administer treatment.
Arm/Group | Upper Arm Treatment With Vacuum Applicator
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.7 [27 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 1
  Caucasian | 24
  Hispanic | 0
  Others | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30
Body Mass Index [Mean (Full Range); unit: kg//m^2] | 28.2 [21.4 to 34.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pre-treatment Images Correctly Identified
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. The review panel will consist of practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Correct identification of photos by at least 2 of the 3 reviewers has an expected success rate of 75%.
Time Frame: 12 weeks post treatment
Population: Thirty subjects received bilateral treatments to the upper arms. Three subjects did not maintain weight per-protocol requirements and were excluded from the primary efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percent correctly identified images
Units Other Than Participants: photo pairs reviewed
Arm/Group | Upper Arm Treatment With Vacuum Applicator
Number analyzed (Participants) | 27
Number analyzed (photo pairs reviewed) | 54
percent correctly identified images | 85.2 [72.9 to 93.4]
Statistical Analysis 1: Comparison: Upper Arm Treatment With Vacuum Applicator; Test type: Other; success proportion = 85.2, 95% CI 2-sided [72.9 to 93.4]

2. Primary Outcome: Safety of the CoolSculpting Device in Upper Arm Treatments
Description: The incidence of reported unanticipated adverse device effects (UADE) from the time of enrollment through the 12-week follow-up visit will be collected and analyzed. It is expected there will be zero UADE's reported.
Time Frame: 12 weeks post-treatment
Population: The analysis population consisted of subjects to whom treatment was administered and who completed the 12 week post-treatment visit.
Measure: Number; unit: UADEs reported
Arm/Group | Upper Arm Treatment With Vacuum Applicator
Number analyzed (Participants) | 30
UADEs reported | 0

ADVERSE EVENTS:
Time Frame: Enrollment through the 12 week follow-up visit.
Arm/Group | Upper Arm Treatment With Vacuum Applicator
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upper Arm Treatment With Vacuum Applicator (N=30)
Prolonged bilateral numbness (Nervous system disorders) | 3 (6) — Four (4) subjects reported prolonged numbness. Bilateral numbness was documented for 3 of the 4 subjects; unilateral numbness was reported for 1 subject.
Tingling outside of treatment area (Nervous system disorders) | 1 (1) — One (1) subject reported minor tingling in the fourth and fifth fingers of one hand immediately after the applicator was removed. The tingling resolved within 20 minutes post-treatment.
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Prolonged unilateral numbness (Skin and subcutaneous tissue disorders) | 1 (1)
Numbness (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach flu (General disorders) | 1 (1)
Cold symptoms (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No